CLINICAL TRIAL: NCT04275271
Title: The Effect of Skill Centered Intervention Based on IMB Model on Promoting School Teachers' Professional Competence in Teaching Sexuality Health
Brief Title: The Effect of Skill Centered Intervention Based on IMB Model on Promoting Teachers' Professional Competence in Teaching Sexuality Health.
Acronym: IMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Mazandaran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IR.TUMS.FNM.REC.1397.102
Record Dates: First submitted 2020-01-06; First posted 2020-02-19 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2019-08

CONDITIONS: Performance
Keywords: skill based intervention,; IMB model,; Professional Competence,; Sexual Health.
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will be received sexuality teaching skills for promotion of professional competence based on information, motivation and behavioral skills model for adolescent sexuality after signing informed consent form and being informed about the goals and details of intervention for 6 sessions (one two hour session per week).
  Interventions: Behavioral: Educational intervention
- Control group (No Intervention): The control group will not receive any intervention until the end of the research.

INTERVENTIONS:
Behavioral: Educational intervention — Skill centered Protocol Training based on IMB model
  Arms: Intervention group

SUMMARY:
Study aim is determining the impact of a skill based intervention based on IMB model on Promoting School Teachers' Professional Competence in Teaching Sexual Health.

DETAILED DESCRIPTION:
This research is a randomized control field trial with two groups; intervention and control. Sampling will be conducted by block design (with block size of 4) random allocation.

Intervention group: Intervention group will be received sexuality teaching skills for promotion of professional competence based on information, motivation and behavioral skills model for adolescent sexuality after signing informed consent form and being informed about the goals and details of intervention for 6 sessions (one two hour session per week).

The control group will not receive any intervention until the end of the research. Then, based on the ethics of the research and their willingness can use the content of program.

ELIGIBILITY:
Inclusion Criteria:

* Having instructors' consent to enter the study, instructor approval for teaching in terms of education system
* Having at least 5 years of teaching experience.

Exclusion Criteria:

* Not participating in at least a third of the sessions
* Not willing to continue cooperation.

Ages: 27 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male teachers who teach in boys' schools
Enrollment: 56 (Estimated)
Dates: Start 2020-04-03 (Estimated); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Changes of mean difference score of professional competence. | Before intervention
  To assess the professional competence of the participants (i.e., knowledge, attitude, skills) by a self-report researcher-made questionnaire.Knowledge and Attitude domain Score from 17 to 85 and Skill Score from 16 to 80. We convert each domain to 0 -100 and report each domain separately and higher scores mean a better outcome
Mean difference score | immediately after the intervention
  To assess the professional competence of the participants (i.e., knowledge, attitude, skills) by a self-report researcher-made questionnaire.Knowledge and Attitude domain Score from 17 to 85 and Skill Score from 16 to 80. We convert each domain to 0 -100 and report each domain separately and higher scores mean a better outcome
Mean difference score | 6 weeks after the intervention
  To assess the professional competence of the participants (i.e., knowledge, attitude, skills) by a self-report researcher-made questionnaire.Knowledge and Attitude domain Score from 17 to 85 and Skill Score from 16 to 80. We convert each domain to 0 -100 and report each domain separately and higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Raziyeh Maasoumi, Assistant, Study Chair — Tehran University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make this available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publishing the results
Access Criteria: Data of the study would be available after unrecognizable process of participants.

REFERENCES:
- [Result] Griewatz J, Simon M, Lammerding-Koeppel M. Competency-based teacher training: A systematic revision of a proven programme in medical didactics. GMS J Med Educ. 2017 Oct 16;34(4):Doc44. doi: 10.3205/zma001121. eCollection 2017. PMID 29085888
- [Result] Defebvre MM, Pavageau M, Chretien A, Carron F, Vanlacken V. [Evaluation of health education training in a French region]. Sante Publique. 2007 Jan-Feb;19(1):39-51. doi: 10.3917/spub.071.0039. French. PMID 17665742
- See also: JSTOR is a not-for-profit service that helps scholars, researchers, and students discover, use, and build upon a wide range of content in a trusted digital archive. We use information technology and tools to increase productivity and facilitate new forms — http://www.jstor.org/page/info/about/policies/terms.jsp